CLINICAL TRIAL: NCT01302184
Title: Robotic Locomotor Experience Applied to Parkinson's Disease (ROLEP)
Brief Title: Robotic Locomotor Experience Applied to Parkinson's Disease
Acronym: ROLEP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Carlo Cisari, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROLEP
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Lokomat®
  Interventions: Device: Lokomat®
- Control Group (Active Comparator): Treadmill training
  Interventions: Device: Treadmill

INTERVENTIONS:
Device: Lokomat® — Patients of the experimental group were trained at 50% of BWS for 15 minutes and 30% of BWS for 15 minutes on the Lokomat®. Treadmill speed was initiated at 1.5km/h and increased to 3.0km/h by increments of 0.5km/h as tolerated.
  A physical therapist supervised the treatment, adjusting treadmill speed and BWS.
  Treatment was performed for 3 days/week, for 4 weeks
  Arms: Experimental Group
Device: Treadmill — Patients of the control group had 30 minutes of treadmill gait training. After having calculated the speed during 6MWT, the patient was trained on a treadmill (RHC770CE - RAM Medical srl). They were trained using 80% of the maximum speed that the patient reached during the test for the first week, 90% for the second week, 100% for the third and fourth week.
  A Physical Therapist provided auditory cueing and direct, continuous feed-back to the patient.
  Treatment was performed for 3 days/week, for 4 weeks.
  Arms: Control Group

SUMMARY:
Gait rehabilitation with treadmill has been reported to be useful in patients with Parkinson's disease. In the last years, interest in robotic devices for gait training has grew up for patients with different neurological disorders, since they minimize demands on physical therapists and may provide a more reliable and constant treatment.

The aim of this study is to evaluate if robotic gait training with Lokomat® can improve walking more than conventional gait training with treadmill in patients affected by Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by PD with a disease stage < III according to Hoehn and Yahr's classification and age < 75 years;
* absence of motor fluctuations;
* able to ambulate independently;
* no treadmill training for at least 6 months before the study.

Exclusion Criteria:

* current levodopa therapy started more than 6 months before enrollment;
* medical or neurological pathology that contributed significantly to gait dysfunction, as musculoskeletal disease, severe osteoarthritis, peripheral neuropathy, previous lower limb joint replacement, cardiovascular disease (recent myocardial infarct, from less than 4 weeks or uncontrolled hypertension, with blood pressure > 180/110 at rest);
* hearth failure (NYHA >=3);
* orthostatic hypotension;
* body weight over 100 kg;
* respiratory disease;
* dementia;
* depression;
* uncorrected visual disturbances.
* patients that have undergone deep brain stimulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
6 minute walking test | Enrollment, after training completion, 3 and 6 months after training completion
  The subject has to walk the longest distance possible within 6 minutes.

SECONDARY OUTCOMES:
10 meter walking test | Enrollment, after training completion, 3 and 6 months after training completion
  The subject has to walk for 16 meters; the maximal speed reached in the central 10 meter is recorded
Time Up and Go test | Enrollment, after training completion, 3 and 6 months after training completion
  The subject has to lift from a chair, walk 3 meters, then turns back and sits on the chair. The time required is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Cisari, MD, Study Director — University of Eastern Piedmont "A. Avogadro" - Dep. Clinical & Experimental Medicine; Stefano Carda, MD, PhD, Principal Investigator — Azienda Ospedaliera-Universitaria "Maggiore della Carità" - Novara
Locations (1):
- Azienda Ospedaliero-Universitaria "Maggiore della Carità", Novara, Italy